CLINICAL TRIAL: NCT06704217
Title: Assessment of the Reliability and Validity of the Six-Spot Step Test in Patients Following Total Hip Arthroplasty
Brief Title: Reliability and Validity of the Six-Spot Step Test After Total Hip Arthroplasty
Acronym: SSST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Elif AYGUN POLAT, PhD, Ordu University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: ODU-SBFTR-AYGUNPOLAT-003; 2024/20 (Other: Ordu University Ethics Committee)
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Total Hip Replacement; Reproducibility of Results; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Other (Experimental): Patients with total hip arthroplasty (THA)
  Interventions: Diagnostic Test: Six Spot Step Test; Diagnostic Test: Oxford Hip Score; Diagnostic Test: Berg Balance Scale

INTERVENTIONS:
Diagnostic Test: Six Spot Step Test — The Six-Spot Step Test (SSST), which evaluates balance and functional ambulation, will be performed in an area 5 meters long and 1 meter wide. Five wooden cylinders will be arranged in a zig-zag pattern within this space, with the last cylinder positioned at the centerline. The participant will be asked to strike the wooden cylinders with the medial or lateral side of the same foot and push them outward. The test will be repeated twice with the dominant foot and twice with the non-dominant foot. A trial will be conducted before the test to familiarize participants with the procedure. A two-minute rest period between the test and trials will be provided to minimize fatigue effects. The test's inter-rater reliability will be assessed by two physiotherapists with more than 5 years of clinical experience, who will administer the test twice at 5-minute intervals.
Diagnostic Test: Oxford Hip Score — The Oxford Hip Score will be used for functional level assessment.
Diagnostic Test: Berg Balance Scale — The Berg Balance Scale (BBS) will be used to assess dynamic balance, which is reliable and commonly used within the orthopedic setting.

SUMMARY:
This study aims to assess the SSST's validity, reliability, and ability to differentiate between high and low fall risk individuals in THA patients. Establishing the SSST as a valid and reliable tool will help manage rehabilitation and apply timely interventions for THA patients.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a common surgery for patients with advanced hip osteoarthritis, aiming to reduce pain and improve function. However, THA patients often experience difficulties in mobility tasks, such as walking, stair climbing, and standing up, even years after surgery. These functional impairments increase the risk of falls, highlighting the need for effective clinical tests to assess balance and mobility. Identifying factors contributing to balance dysfunction and implementing appropriate rehabilitation are crucial for improving quality of life.

The Six-Spot Step Test (SSST), developed by Nieuwenhuis et al., is a quick and easy test that evaluates balance and mobility in daily life activities. However, its validity and reliability in THA patients have not been studied. This research aims to assess the SSST's validity, reliability, and ability to differentiate between high and low fall risk individuals in THA patients. Establishing the SSST as a valid and reliable tool will help manage rehabilitation and apply timely interventions for THA patients.

ELIGIBILITY:
Inclusion Criteria:

* Underwent primary unilateral Total Hip Arthroplasty (THA)
* Surgery performed using the posterolateral approach
* At least six months of postoperative follow-up

Exclusion Criteria:

* Patients who underwent bilateral or revision THA
* History of additional lower limb surgery
* Body mass index (BMI) greater than 40 kg/m²
* Neurological, orthopedic, or systemic disorders that could impair gait or balance

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Six Spot Step Test-1 | Day 1
  The SSST wil be measured by the first investigator
Six Spot Step Test-2 | Day 1
  The SSST wil be measured by the second investigator
Six Spot Step Test-3 | 7-10 days after
  The SSST wil be measured by the first investigator
Six Spot Step Test-4 | 7-10 days after
  The SSST wil be measured by the second investigator
Timed Up and Go test | Day 1
  A timed up and go test test will be measured for validity analysis.
Four Square Step Test | Day 1
  A four square step test will be measured for validity analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Elif AYGUN POLAT, PhD, Study Director — Ordu University; Yusuf POLAT, Assoc. Prof., Principal Investigator — Ordu University; Sevim ACAROZ, Assoc. Prof., Principal Investigator — Ordu University; Yunus Emre OZBILEN, MD, Principal Investigator — Ordu University; Alper ÇIRAKLI, Prof., Study Chair — Ordu University
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Aygun-Polat E, Polat Y, Ozbilen YE, Altun A, Acaroz S, Cirakli A. Reliability and validity of the Six-Spot Step Test in patients with total hip arthroplasty. Physiotherapy. 2026 Mar;130:101848. doi: 10.1016/j.physio.2025.101848. Epub 2025 Sep 15. PMID 41289866